CLINICAL TRIAL: NCT02928835
Title: Effects of Dynamic Splinting on Knee Flexion Angle After Total Knee Arthroplasty: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Eros de Oliveira Jr, Principal Investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ethical Protocol n°: 11.049
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Acquired Fixed Flexion Deformity of the Knee (Disorder)
Keywords: Total knee arthroplasty; Knee flexion; Dynamic orthosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynasplint group (Experimental): The experimental group received standardized physical therapy intervention and used the knee flexion Dynasplint orthosis six hours daily during one month, starting at day seven after total knee arthroplasty surgery.
  Interventions: Device: Knee flexion Dynasplint orthosis
- Control group (No Intervention): Control group received standardized physical therapy intervention.

INTERVENTIONS:
Device: Knee flexion Dynasplint orthosis — Standardized rehabilitation procedures started at the first day after total knee arthroplasty. Both groups received the same standardized physical therapy intervention. The experimental group used the knee flexion Dynasplint orthosis (Dynasplint Systems, Inc. Canada, Woodbridge, ON) at night, while sleeping, over six continuous hours for one month, starting seven days after the total knee arthroplasty. The control group received only the standardized physical therapy intervention.
  Other Names: Dynasplint
  Arms: Dynasplint group

SUMMARY:
To evaluate the effects of a knee flexion Dynasplint orthosis on knee flexion angle after a total knee arthroplasty. Sixty participants, who underwent a total knee arthroplasty, were randomly assigned in two groups: control group and Dynasplint group.

DETAILED DESCRIPTION:
Post-surgical rehabilitation interventions following total knee arthroplasty consist mainly of stretching exercises to improve flexibility and prevent soft tissue fibroses around the joint, thus, avoiding contractures and providing increases in the range of motion at the knee joint. Although knee manipulation and open arthrolysis may improve range of motion after total knee arthroplasty , the results have been variable and additional procedures are frequently necessary. Studies demonstrated the effectiveness of dynamic orthoses in reducing joint contractures after orthopedic surgeries in various joints that require a long rehabilitation period. Therefore, the purpose of the present study was to evaluate the effects of the knee flexion Dynasplint orthosis (KFD) on the length of rehabilitation and range of knee flexion angle after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled will have been schedule to receive first prosthesis of the knee:

Arthritis of the knee, dominated with pain Painful, deformed, and/or unstable knees secondary to degenerative or inflammatory conditions

Exclusion Criteria:

Fractures Knee sepsis Osteomyelitis or any orthopedic infection Psoriasis Knee joint neuropathy Previous Stroke or Brain Injury Significant pathology acquired secondary to the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The knee flexion angle was assessed in supine position with a universal goniometer | Change from baseline knee flexion angle at 6 months
  The outcomes were obtained by one experienced and well-trained physical therapist.

SECONDARY OUTCOMES:
Measures of knee function. | Change from baseline knee flexion angle at 6 months
  Assessed by the Knee Society Score (KSS)
Measures for quality of life | Change from baseline knee flexion angle at 6 months
  Assessed by Short-form 36 Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Eros De Oliveira Jr, PhD, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Hôpital Jean-Talon, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nadler SF, Malanga GA, Zimmerman JR. Continuous passive motion in the rehabilitation setting. A retrospective study. Am J Phys Med Rehabil. 1993 Jun;72(3):162-5. doi: 10.1097/00002060-199306000-00011. PMID 8512680
- [Background] Meier W, Mizner RL, Marcus RL, Dibble LE, Peters C, Lastayo PC. Total knee arthroplasty: muscle impairments, functional limitations, and recommended rehabilitation approaches. J Orthop Sports Phys Ther. 2008 May;38(5):246-56. doi: 10.2519/jospt.2008.2715. Epub 2007 Dec 14. PMID 18448878
- [Background] Shakespeare D, Kinzel V. Rehabilitation after total knee replacement: time to go home? Knee. 2005 Jun;12(3):185-9. doi: 10.1016/j.knee.2004.06.007. No abstract available. PMID 15911290
- [Background] Kotani A, Yonekura A, Bourne RB. Factors influencing range of motion after contemporary total knee arthroplasty. J Arthroplasty. 2005 Oct;20(7):850-6. doi: 10.1016/j.arth.2004.12.051. PMID 16230234
- [Background] Miner AL, Lingard EA, Wright EA, Sledge CB, Katz JN; Kinemax Outcomes Group. Knee range of motion after total knee arthroplasty: how important is this as an outcome measure? J Arthroplasty. 2003 Apr;18(3):286-94. doi: 10.1054/arth.2003.50046. PMID 12728419
- [Background] Furia JP, Willis FB, Shanmugam R, Curran SA. Systematic review of contracture reduction in the lower extremity with dynamic splinting. Adv Ther. 2013 Aug;30(8):763-70. doi: 10.1007/s12325-013-0052-1. Epub 2013 Sep 10. PMID 24018464
- [Background] Gaspar PD, Willis FB. Adhesive capsulitis and dynamic splinting: a controlled, cohort study. BMC Musculoskelet Disord. 2009 Sep 7;10:111. doi: 10.1186/1471-2474-10-111. PMID 19735563
- [Background] Finger E, Willis FB. Dynamic splinting for knee flexion contracture following total knee arthroplasty: a case report. Cases J. 2008 Dec 29;1(1):421. doi: 10.1186/1757-1626-1-421. PMID 19113998
- [Background] Farahini H, Moghtadaei M, Bagheri A, Akbarian E. Factors influencing range of motion after total knee arthroplasty. Iran Red Crescent Med J. 2012 Jul;14(7):417-21. Epub 2012 Jul 30. PMID 22997557
- [Background] Kucera T, Urban K, Karpas K, Sponer P. [Restricted motion after total knee arthroplasty]. Acta Chir Orthop Traumatol Cech. 2007 Oct;74(5):326-31. Czech. PMID 18001629
- [Background] Denis M, Moffet H, Caron F, Ouellet D, Paquet J, Nolet L. Effectiveness of continuous passive motion and conventional physical therapy after total knee arthroplasty: a randomized clinical trial. Phys Ther. 2006 Feb;86(2):174-85. PMID 16445331
- [Background] Ritter MA, Harty LD, Davis KE, Meding JB, Berend ME. Predicting range of motion after total knee arthroplasty. Clustering, log-linear regression, and regression tree analysis. J Bone Joint Surg Am. 2003 Jul;85(7):1278-85. doi: 10.2106/00004623-200307000-00014. PMID 12851353
- [Background] MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW, Kramer J, Vaz M. Prospective randomized clinical trial of continuous passive motion after total knee arthroplasty. Clin Orthop Relat Res. 2000 Nov;(380):30-5. doi: 10.1097/00003086-200011000-00005. PMID 11064970
- [Background] Beaupre LA, Davies DM, Jones CA, Cinats JG. Exercise combined with continuous passive motion or slider board therapy compared with exercise only: a randomized controlled trial of patients following total knee arthroplasty. Phys Ther. 2001 Apr;81(4):1029-37. PMID 11296803